CLINICAL TRIAL: NCT03372382
Title: Ibuprofen and Acetaminophen Versus Ibuprofen and Acetaminophen Plus Hydrocodone for Analgesia After Cesarean Section: A Prospective, Randomized Control Trial
Brief Title: Ibuprofen and Acetaminophen Versus Ibuprofen and Acetaminophen Plus Hydrocodone for Analgesia After Cesarean Section
Acronym: IVY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jenifer Dinis Ballestas, MD, Maternal Fetal Medicine Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-17-0777
Record Dates: First submitted 2017-12-09; First posted 2017-12-13 (Actual); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Opioid Use; Pain, Postoperative
Keywords: postpartum
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Acetaminophen; oxycodone-acetaminophen

STUDY DESIGN:
Intervention Model Description: two parallel groups included, randomized to control analgesic regimen versus alternative analgesic regimen and followed prospectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ibuprofen plus acetaminophen (Active Comparator): women that had a C-section will be discharged home with prescriptions for ibuprofen and acetaminophen
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen
- ibuprofen plus acetaminophen/hydrocodone (Experimental): women that had a C-section will be discharged home with prescriptions for ibuprofen and acetaminophen/hydrocodone (Norco)
  Interventions: Drug: Ibuprofen; Drug: Norco

INTERVENTIONS:
Drug: Ibuprofen — NSAID
Drug: Acetaminophen — analgesic
  Arms: ibuprofen plus acetaminophen
Drug: Norco — acetaminophen plus opioid
  Arms: ibuprofen plus acetaminophen/hydrocodone

SUMMARY:
Postpartum patients delivered by cesarean section will be randomized to NSAIDS Vs NSAIDS plus opioid

DETAILED DESCRIPTION:
Women will be approached priors to discharge from the hospital, if they meet inclusion criteria and consent for the study, they will be randomized to one of two possible analgesic regimens. They will be followed at 1-2 weeks and 4-6 weeks after discharge to assess pain level.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaker women who had a cesarean section

Exclusion Criteria:

* Inability or refusal to provide informed consent.
* Reported current or prior opioid or benzodiazepine use disorder, including urine drug screen positive for a non prescribed opioid or benzodiazepine upon admission or during prenatal care.
* Current treatment with methadone, buprenorphine or buprenorphine plus naloxone.
* Known alcoholism disorder.
* Severe renal or hepatic impairment.
* Known creatinine > 1.5 at the time of delivery or severe proteinuria leading to diagnosis of renal disease prior to delivery.
* Severe peptic ulcer disease
* Severe asthma (if patient has asthma but has previously tolerated NSAIDS, she will be allowed to participate)
* Known CYP450/CY92D6 mutation conferring opioid ultra-rapid metabolizer status.
* Allergy to any of the study drugs (anaphylaxis).
* Incarcerated or institutionalized patients.
* Inability to follow up as outpatient in our outpatient clinic.
* wound dehiscence or infection diagnosed prior to discharge from the hospital
* wound vac placed prior to discharge from the hospital

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — study will be conducted among subjects who delivered by cesarean section, which by definition, are only females.
Enrollment: 170 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenifer Dinis, MD, Principal Investigator — UT Houston, McGovern Medical School
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment start date: 12/2017 recruitment end date: 03/2018
Groups:
- Ibuprofen Plus Acetaminophen: women that had a C-section will be discharged home with prescriptions for ibuprofen and acetaminophen
  Ibuprofen: NSAID
  Acetaminophen: analgesic
  85 women recruited into this study arm
- Ibuprofen Plus Acetaminophen/Hydrocodone: women that had a C-section will be discharged home with prescriptions for ibuprofen and acetaminophen/hydrocodone
  Ibuprofen: NSAID
  Acetaminophen plus hydrocodone: Opioid
  85 women recruited into this study arm
Period: Overall Study
Arm/Group | Ibuprofen Plus Acetaminophen | Ibuprofen Plus Acetaminophen/Hydrocodone
Started | 85 | 85
Completed | 76 | 81
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen Plus Acetaminophen | Ibuprofen Plus Acetaminophen/Hydrocodone | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.39 (5.8) | 28.05 (5.64) | 28.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 85 | 170
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African american | 36 | 49 | 85
  Race: Hispanic | 34 | 29 | 63
  Race: white | 13 | 3 | 16
  Race: other | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pain Level
Description: pain level measured by objective and subjective scales.
  1- Objective scale: visual analogue pain score (VAS). It is a 100 mm line, patients will be instructed to mark a point in the line that represents their pain level. A point towards the left will mean "less pain" and a point towards the right will mean "more pain". After the patient makes a selection, the research team will measure where the selected point is (in cm). minimum measurement =0mm = no pain. maximum measurement=100mm=worst pain.
Time Frame: 2-4 weeks postpartum
Population: The primary outcome was available in 71 patients in the non-opioid group and 76 patients in the opioid group. The results below are primary outcome data analyzed by intention to treat.
Measure: Mean (Standard Deviation); unit: millimeters on a scale
Arm/Group | Ibuprofen Plus Acetaminophen | Ibuprofen Plus Acetaminophen/Hydrocodone
Number analyzed (Participants) | 71 | 76
millimeters on a scale | 12.3 (19.5) | 15.9 (20.4)
Statistical Analysis 1: Comparison: Ibuprofen Plus Acetaminophen vs Ibuprofen Plus Acetaminophen/Hydrocodone; Sample size calculations were based on VAS pain score at 2-4 weeks, assuming a mean of 10mm and standard deviation (SD) of 20 mm in the opioid group Assuming a two-sided alpha level of 0.05 and 80% power to detect equivalence, a total of 138 participants would be needed. To account for a 25% expected attrition rate and crossover, a total of 170 participants would be needed; Test type: Equivalence — We prespecified an equivalence margin of -10 to 10mm. We would consider non-opioid analgesia to be equivalent to opioid analgesia if the pain score mean difference between the groups and it's 95% confidence interval (CI) were within the prespecified margin. Pain score mean difference or 95% CI boundaries outside this range would be considered a clinically important difference between treatments; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-2.1 to 11.9] — The upper boundary of the CI is out of pre-specified limits

2. Secondary Outcome: Patient Satisfaction
Description: patient satisfaction as measured by the following scale: 1(very dissatisfied) 2(somewhat dissatisfied) 3(neutral) 4(satisfied) 5(very satisfied)
Time Frame: 2-4 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen Plus Acetaminophen | Ibuprofen Plus Acetaminophen/Hydrocodone
Number analyzed (Participants) | 76 | 81
Participants
  1(very dissatisfied) | 2 | 4
  2(somewhat dissatisfied) | 3 | 3
  3(neutral) | 11 | 12
  4(satisfied) | 23 | 16
  5(very satisfied) | 37 | 46

ADVERSE EVENTS:
Time Frame: four months
Description: a standard questionnaire was used to assess whether any adverse events had occurred. It was administered at the time of follow up.
  Medical records were also reviewed to determine if a patient had an adverse event
Arm/Group | Ibuprofen Plus Acetaminophen | Ibuprofen Plus Acetaminophen/Hydrocodone
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 14/85 | 25/85
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen Plus Acetaminophen (N=85) | Ibuprofen Plus Acetaminophen/Hydrocodone (N=85)
nausea / emesis (Gastrointestinal disorders) | 2 (2) | 4 (5) — non-opioid group: 2 opioid group: 5
constipation (Gastrointestinal disorders) | 7 (7) | 13 (13) — constipation
somnolence (General disorders) | 4 (4) | 13 (13) — somnolence
GERD (Gastrointestinal disorders) | 1 (1) | 2 (2) — reflux
itching (General disorders) | 1 (1) | 2 (2) — itching

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT03372382/Prot_SAP_000.pdf